CLINICAL TRIAL: NCT01709591
Title: Effect of Targeted Prenatal Education on Perceptions of Epidural on Acceptance of Epidural Analgesia: a Randomized Controlled Trial
Brief Title: Effect of Prenatal Education on Perceptions of Epidural Acceptance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Santa Clara Valley Health & Hospital System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-081
Record Dates: First submitted 2012-10-15; First posted 2012-10-18 (Estimated); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Labor Pain
Keywords: intrapartum pain management, epidural
MeSH Terms: conditions — Labor Pain | interventions — Prenatal Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- No Prenatal education (No Intervention): These subjects will be randomized to receive routine prenatal epidural class (control group).
- Receives Prenatal Education (Active Comparator): Subjects randomized to this group will receive educational video addressing the cultural and perceptions regarding the myths on epidural in either English or Spanish (Keeping an Open Mind: choices in Labor Anaglesia: an educational produce of the Society for Obstetric Anesthesia and perinatology)
  Interventions: Behavioral: Prenatal education

INTERVENTIONS:
Behavioral: Prenatal education
  Arms: Receives Prenatal Education

SUMMARY:
The purpose of the study is to determine if targeted prenatal educational program on womens' perceptions of epidural increases the acceptance of intrapartum epidural analgesia relative to the control group.

DETAILED DESCRIPTION:
Racial/ethnic disparities exist in the proportion of patients receiving epidural analgesia. The purpose of our study is to determine if culturally-sensitive educational program targeting womens' perceptions of epidural increases the acceptance of intrapartum epidural use.

ELIGIBILITY:
Inclusion Criteria:

1. Women with viable intrauterine gestation seeking prenatal care
2. Candidates for Intrapartum epidural analgesia

Exclusion Criteria:

1. Intrapartum epidural analgesia is contraindicated
2. Trial of labor is contraindicated.
3. Patients planning an elective cesarean

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 111 (Actual)
Dates: Start 2011-06; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
pre and post intervention PEQ survey results to elucidate the changes in perceptions of epiduralepidural based on the PEQ survey | One year time period
  All subjects will be asked to fill out the Perceptions on Epidural Questionnaire (PEQ) to elucidate their desire to receive intrapartum pain control & their attitude towards epidural to patients. Each survey will take approximately five to ten minutes to complete. The survey will be distributed in English and Spanish.

CONTACTS AND LOCATIONS:
Overall Officials: Anita Sit, MD, Principal Investigator — Santa Clara Valley Health and Hospital System
Locations (1):
- Santa Clara Valley Health and Hospital System, San Jose, California, United States